CLINICAL TRIAL: NCT05010213
Title: The Effect of Training Given With the Roy Adaptation Model on the Self-care Agency and Coping Strategies of Patients With Plaster Casts.
Brief Title: Plaster Patient Education With Roy Adaptation Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Nida AYDIN, Research assistant, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NAYDIN
Record Dates: First submitted 2021-07-29; First posted 2021-08-18 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Educational Problems
Keywords: Coping Skills; Casts, Surgical; Patient Education as Topic; Nursing Education; Self Care
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): There will be no intervention to the control group.
- Experimental group (Experimental): The experimental group will be given training based on the roy adaptation model.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Educational intervention
  Arms: Experimental group

SUMMARY:
The aim of this study is to determine the effect of training given with the Roy adaptation model on the self-care agency and coping strategies of patients with plaster casts.

DETAILED DESCRIPTION:
According to Global Burden of Disease data, fractures, which 436 million people suffer from each year, are the second most common musculoskeletal system disorder. Plaster casts have been used in treatment of fractures since 1850, and they play an important role in extremity injuries and the healing of operative repairs. In fractures treated with plaster, the bone alignment is corrected and this alignment is maintained with limited mobility. However, if plaster casts are incorrectly applied or not properly taken care of, this may prevent the healing of fractures and can threaten the safety of patients. Failure to comply with plaster-casting and cast-care principles can cause patients a range of immediate and delayed complications, including severe pain, edema, compartment syndrome, tissue necrosis, malunion, delayed union, nonunion, contracture, neurological problems, paralysis and pressure sores. Orthopedic patients, and especially those with plaster casts, are susceptible to the side effects arising from immobility. They thus need quality care and information to prevent or manage these side effects. Nurses play an important role in prevention or early recognition of complications arising from plaster-casting and in providing the patient with information. Orthopedic nursing requires special skills, knowledge and clinical judgement to provide the plaster cast-patient with safe, quality-care and to prevent complications. Patient education and information are very important for those patients whose treatment continues at home after casting, in order that they can maintain their care and prevent complications.In this study, the sample size was determined with an effect size of 0.43 using the power analysis Gpower 3.1.9.7 program. Accordingly, it was calculated that 29 patients were included in the intervention and control groups with a 5% margin of error and 80% power. İt was decided to include at least 66 people in each working group with 10% surplus, considering that they might be lost in data collection.

ELIGIBILITY:
Inclusion Criteria:

* With lower extremity fracture
* Have at least 6 weeks of plaster cast experience

Exclusion Criteria:

* Have communication problem
* Have restriction of movement before fracture
* Patient who can not speak very well Turkish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-12-08 (Actual)

PRIMARY OUTCOMES:
Self-care agency scale score level | At the beginning of plaster treatment, an avarage of 1 hour
  Score level of self-care agency before the patient education
Coping orientation to problems experienced (COPE) | At the beginning of plaster treatment, an avarage of 1 hour
  Score level of coping orientation to problems experienced before the patient education

SECONDARY OUTCOMES:
Self-care agency scale score level | At the end of treatment, an avarage of 1 week
  Score level of coping orientation to problems experienced after the patient education
Coping orientation to problems experienced (COPE) | At the end of treatment, an avarage of 1 week
  Score level of coping orientation to problems experienced after the patient education

CONTACTS AND LOCATIONS:
Locations (1):
- Near East University, Nicosia, Cyprus